CLINICAL TRIAL: NCT02014012
Title: Evaluation of Pulse Wave Velocity as a Predictive Factor for Postoperative Cardiovascular Complication After Cardiac Surgery: a Prospective Study
Brief Title: PWV for Cardiovascular Complication After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jae-Sung Choi, MD. PhD., Associate Professor, Seoul National University Hospital
Other Study IDs: 16-2013-40; PWV-OHS (Other: SMG-SNU Boramae Medical Center)
Record Dates: First submitted 2013-07-31; First posted 2013-12-17 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: C.Surgical Procedure; Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Arterial stiffness has been suggested as an independent risk factor for the development of coronary artery disease and stroke. Pulse wave velocity (PWV) is an noninvasive established index to quantify arterial stiffness. Therefore, we try to investigate the correlation between PWV values and cardiovascular complications like stroke, acute renal failure, or perioperative myocardial infarction after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery patients who sign the informed consent

Exclusion Criteria:

* Chronic renal failure (Cr>1.5mg/dL), Dialysis patients
* Previous stroke
* Left ventricular dysfunction (EF <50%)
* ASO with claudication
* < 40 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Postoperative cardiovascular complication and parameters | within the first 7 days after surgery
  Stroke, Delirium, Newly developed atrial fibrillation, ARF, Peak CK-MB and troponin I levels measured at 12 and 24 hours after surgery, Peak estimated GFR and corresponding creatinine

SECONDARY OUTCOMES:
E/e' and e' measured by transthoracic echocardiography with color-coded tissue dopper imaging in patients undergoing non-valvular cardiac surgery | baseline and within the first 14 days after surgery
  peak early transmitral filling velocity during early diastole (E), mean early velocity at the septal mitral annulus (e')

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea